CLINICAL TRIAL: NCT05047159
Title: Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Brief Title: The Role of Neuromodulation Technique In Depression Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-74
Record Dates: First submitted 2021-08-09; First posted 2021-09-16 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Phototherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- drug therapy group (Experimental): Drug: drug therapy There is no restriction on the choice of therapeutic drugs.
  Interventions: Drug: drug therapy
- drug therapy combined with repetitive transcranial magnetic stimulation (rTMS) group (Experimental): Device: rTMS Stimulation will be performed for 20 working days once a day (4 weeks). Extend course to 30 sessions (6 weeks) in responders who have not achieved symptom remission.
  Frequency: 10Hz; Intensity: 110% RMT; Coil-type: F8; Sessions-pulse: 3000; Site: the left dorsolateral prefrontal cortex.
  Drug: drug therapy There is no restriction on the choice of therapeutic drugs.
  Interventions: Device: rTMS; Drug: drug therapy
- drug therapy combined with light therapy group (Experimental): Device: light therapy Active 10,000-lux fluorescent white light box for 30 min/d in the early morning for 6 weeks.
  Drug: drug therapy There is no restriction on the choice of therapeutic drugs.
  Interventions: Device: light therapy; Drug: drug therapy
- drug therapy combined with electroconvulsive therapy (ECT) group (Experimental): Device: ECT The electrode placements are bifrontal (BF); the electrical intensity is 1.5 to 2.0 times the seizure threshold (ST); 3 times per week.
  Drug: drug therapy There is no restriction on the choice of therapeutic drugs.
  Interventions: Device: ECT; Drug: drug therapy
- drug therapy combined with magnetic seizure therapy (MST) group (Experimental): Device: MST A coil placement at the vertex (i.e., Cz in 10-20 electroencephalogram [EEG] system) with a frequency of stimulation of 100 Hz, pulse width of 0.2 to 0.4 ms, and stimulation duration of 10 seconds; 2 times per week.
  Drug: drug therapy There is no restriction on the choice of therapeutic drugs.
  Interventions: Device: MST; Drug: drug therapy

INTERVENTIONS:
Device: rTMS — Stimulation will be performed for 20 working days once a day (4 weeks). Extend course to 30 sessions (6 weeks) in responders who have not achieved symptom remission.
  Frequency: 10Hz; Intensity: 110% RMT; Coil-type: F8; Sessions-pulse: 3000; Site: the left dorsolateral prefrontal cortex.
  Arms: drug therapy combined with repetitive transcranial magnetic stimulation (rTMS) group
Device: light therapy — Active 10,000-lux fluorescent white light box for 30 min/d in the early morning for 6 weeks.
  Arms: drug therapy combined with light therapy group
Device: ECT — The electrode placements are bifrontal (BF); the electrical intensity is 1.5 to 2.0 times the seizure threshold (ST); 3 times per week.
  Arms: drug therapy combined with electroconvulsive therapy (ECT) group
Device: MST — A coil placement at the vertex (i.e., Cz in 10-20 electroencephalogram [EEG] system) with a frequency of stimulation of 100 Hz, pulse width of 0.2 to 0.4 ms, and stimulation duration of 10 seconds; 2 times per week.
  Arms: drug therapy combined with magnetic seizure therapy (MST) group
Drug: drug therapy — There is no restriction on the choice of therapeutic drugs.

SUMMARY:
This study aims to explore the efficacy, safety and long-term effects of common and available non-invasive neuromodulation techniques in the treatment of depression, and to provide a data basis for the establishment of individualized treatment and efficacy prediction models. 450 patients will be enrolled and randomly assigned to five different treatments. Psychopathological assessment will be performed in both acute and maintenance phases of treatment with the Hamilton Depression Rating Scale, the Hamilton Anxiety Rating Scale, and the Patient Health Questionaire-9, the Sheehan Disability Scale, the Vascular Quality of Life-6 Questionnaire respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60;
2. Meet the DSM-IV "major Depressive Episode" diagnostic criteria and are currently in the depressive episode (MDE) stage;
3. The 17-item Hamilton Depression Scale (HAMD-17) score was > 17, and the HAMD-17 item 1 (depression) score was ≥2;
4. Failure to respond adequately to at least one of the new antidepressants (including a HAMD-17 reduction rate of less than 50% and an intolerant drug side effect);
5. Junior high school education or above, with sufficient audio-visual understanding of the research content, and signed the informed consent;
6. If drug therapy is used at the same time, the medication regimen should remain unchanged at least 4 weeks before the follow-up group, and continue to remain unchanged during the neurological intervention in the acute phase;
7. Right-handed.

Exclusion Criteria:

1. Schizophrenia, or psychotic symptoms unrelated to depression, bipolar disorder, eating disorder, etc.;Personality disorders and mental retardation;Patients with depression caused by physical diseases;
2. Suffering from the following serious diseases:History of brain injury or cerebrovascular accident, narrow-angle glaucoma, epilepsy, myocardial infarction, unstable angina pectoris, congestive heart failure, severe cirrhosis, acute and chronic renal failure, severe diabetes, aplastic anemia,Moderate to severe malnutrition and other serious neurological, heart, liver, kidney, endocrine, blood system and other physical diseases or diseases that may interfere with the study (abnormal index is more than 2 times the normal value);
3. Patients with metal implants or electronic instruments (such as embedded intracranial electrodes, cochlea, medical pump, etc.), photosensitive dermatitis and other skin diseases or other contraindications in the body;
4. Intracranial mass, cerebral infarction, increased intracranial pressure, or other active central nervous system disease, including epilepsy;Dementia, delirium, memory loss or other cognitive disorders;Brain trauma that increases the risk of seizures;
5. Severe drug allergic reaction;
6. Pregnant, lactating or planning to become pregnant;
7. Substance abuse (excluding caffeine and nicotine) in the past 3 months;
8. Received rTMS, tDCS, tACS, light therapy, ECT, MST, DBS therapy in the past 3 months;
9. Serious suicide attempt (hamD-17 item 3 "suicide" score ≥3);
10. Refuse to sign the informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the change of the HAMD-17 score | baseline, and 1, 2, 4, 8, 12, 24, 36, 48 weeks.
  the change of HAMD-17 score between baseline and after treatment.

SECONDARY OUTCOMES:
remission rate | 12, 24, 36, 48 weeks.
  HAMD-17 total score ≤ 7 after treatment.
response rate | 12, 24, 36, 48 weeks.
  a reduction rate of HAMD-17 score ≥ 50% from baseline after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No